CLINICAL TRIAL: NCT00175695
Title: A Safety and Efficacy Trial of Recombinant Human Activated Protein C in Both Early-onset Pre-eclampsia and Severe Postpartum Pre-eclampsia.
Brief Title: Disease Modification in Toxaemia of Pregnancy
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Peter von Dadelszen, University of British Columbia
Other Study IDs: C03-0230; F1K-CA-0013; 9427-C2266-22C
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-02-04 (Estimated); Status verified 2011-02

CONDITIONS: Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — drotrecogin alfa activated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Recombinant human activated protein C or drotrecogin alpha — We are going to investigate a compound (recombinant human activated protein C (rhAPC)) that has the potential to modify disease activity in pre-eclampsia by reducing coagulation and inflammation disorders.

SUMMARY:
Short description of the primary purpose of the protocol intended for the lay public. Include brief statement of study hypothesis

Pre-eclampsia (toxemia of pregnancy) is the most cause of death among pregnant women in North America. It also causes many complications for fetuses (unborn children) and neonates (newborn children). Pre-eclampsia is defined by high blood pressure (hypertension), the loss of protein into the urine (proteinuria), and disorders of many body systems, including the blood clotting (coagulation) and inflammation. What is needed is a compound that will safely prolong pregnancies, to give babies more time to grow inside their mothers, and will help the recovery in those mothers after delivery.

We are going to investigate a compound (recombinant human activated protein C (rhAPC)) that has the potential to modify disease activity in pre-eclampsia by reducing coagulation and inflammation disorders. rhAPC is effective in patients suffering from septic shock. We will test rhAPC in women who develop severe pre-eclampsia in two ways. First, in women with severe pre-eclampsia remote from term who are carrying small babies (intent: safely prolong their pregnancies). Second, in women who have had severe pre-eclampsia before their baby delivered (including women in the first group), or whose disease develops/worsens after delivery (intent: switch off the disease so dangerous complications do not arise).

This study is a preliminary one to look for possible risks and benefits for these women. Only 40 women will be studied to provide initial evidence on which to base a larger international trial which is planned. We will study their pregnancy outcomes as well as markers of disease activity, to gain a better understanding of the mechanisms by which these women become unwell.

ELIGIBILITY:
Inclusion Criteria:

* Scenario 1 is severe early-onset pre-eclampsia, where the fetal prognosis is dismal (<50% chance of intact survival [disease onset <27+0 weeks gestation and/or estimated fetal weight <600g].
* Scenario 2 is postpartum pre-eclampsia, where there is either severe antenatal disease, deteriorating postpartum disease, or de novo postpartum disease.

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with pre-eclampsia ('toxaemia of pregnancy').
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Antenatal: The primary safety outcome will be the incidence of peripartum bleeding, The primary efficacy outcome will be days of pregnancy prolongation | Unknown at this time
Postnatal: The primary safety outcome will be the incidence of postpartum bleeding. The primary efficacy outcome will be 'days alive and free of illness' | Unknown at this time

SECONDARY OUTCOMES:
We will assess disease activity (as measured by clinical and basic science indices). | Unknown at this time

CONTACTS AND LOCATIONS:
Overall Officials: Peter von Dadelszen, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital and Health Centre, Vancouver, British Columbia, Canada